CLINICAL TRIAL: NCT04737954
Title: A Performance Evaluation of the LumiraDx Point Of Care D-dimer Assay
Acronym: EMBOL1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00006
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: IVD Performance Evaluation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected VTE patients (Experimental): Venous blood draw of up to 20ML and up to 6 fingerstick capillary draws
  Interventions: Diagnostic Test: Venepuncture; Diagnostic Test: Fingerstick

INTERVENTIONS:
Diagnostic Test: Venepuncture — Venous blood draw
Diagnostic Test: Fingerstick — Capillary blood draw

SUMMARY:
In patients with symptoms of Venous Thromboembolism (VTE) (mainly deep vein thrombosis (DVT) or pulmonary embolism (PE)), the study will evaluate the agreement between the D-Dimer measurements from the LumiraDx POC D-Dimer assay and a reference method, as an aid in diagnosis, assessment and exclusion of DVT and PE.

DETAILED DESCRIPTION:
This is a performance evaluation study designed to assess the precision and accuracy of the LumiraDx Point of Care (POC) D-Dimer test when used in patients presenting with symptoms of Venous thromboembolism (VTE), which mainly comprises deep vein thrombosis (DVT) or pulmonary embolism (PE).

The LumiraDx POC D-Dimer test is a quantitative immunoassay providing results in under 10 minutes. The accuracy of the LumiraDx POC D-Dimer test will be assessed using capillary whole blood, venous blood, and plasma samples, by comparison to the D-Dimer results obtained from the same individuals as analysed by trained laboratory professionals using a reference device. The results of this study are intended to be used for regulatory filings for use as an in vitro diagnostic test in the European Union (EU) and other relevant geographies.

Adult males and females presenting to the study sites with symptoms of VTE will be included in the study. Approximately 1000 subjects will be recruited in total. An initial analysis will be completed on the first 200 patients to determine accuracy of the LumiraDx D-Dimer test versus the reference method. The study will continue until 1000 patients are recruited and with a minimum of 120 confirmed VTE events, in order to complete retrospective analysis using the LumiraDx D-Dimer cut-off for exclusion of VTE.

Once consent is obtained, blood tube samples will be drawn and finger-stick samples of capillary blood will be taken from the subject, these will be applied directly to unique test strips for immediate measurement of D-Dimer on the LumiraDx POC D-Dimer test.

The D-Dimer results obtained via the LumiraDx D-Dimer test will be used in a set of comparative analyses designed to determine the performance characteristics of the test. This study is an observational, cross-sectional design. As an observational study of an investigative device, results obtained during the course of the study will not inform or alter patient management or treatment decisions in any way.

ELIGIBILITY:
Inclusion Criteria:

Subject is greater or equal to 18 years of age Willing and able to provide written informed consent and comply with study procedures Symptoms of thromboembolic event

Exclusion Criteria:

Suspected Sinus Venous Thromboembolism / Cerebral Venous Sinus Thromboembolism End-stage renal failure on haemodialysis Current anticoagulant therapy (Fragmin, LMWH) within the last 30 days Patient has previously participated in this study Life expectancy documented as <30 days Haemodynamically unstable (e.g. cardiogenic shock) Patients taking anticoagulant therapy (DOACS, Warfarin, Heparins etc) within the last 30 days Patient deemed medically unfit to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Determine the accuracy of the LumiraDx POC D-Dimer assay when compared to a reference method in patients with suspected VTE. | 2 months
  Measurement of blood samples from patients with suspected VTE in a reference method and in the LumiraDx method to assess accuracy of the LumiraDx method.
Assessment of accuracy of using the D-Dimer cut-off set by the LumiraDx D-Dimer test in excluding patients with symptoms of VTE (DVT and PE) when used in combination with the pre-probability test (Wells Score). | 10 months
  Measurement of blood samples from patients with suspected VTE in the LumiraDx D-dimer assay in conjunction with pre-test probability score and final clinical outcome in order to set a clinical cut-off for the LumiraDx D-dimer assay

CONTACTS AND LOCATIONS:
Overall Officials: Richard Body, Principal Investigator — Professor of Emergency Medicine
Locations (13):
- Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg, Germany
- United Kingdom (12):
  - Addenbrookes Hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Epsom and St Helier Hospitals, Epsom
  - Glsagow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - St Johns Hospital, Livingston
  - Homerton University Hospital NHS Foundation Trust, London
  - Royal London Hospital, London
  - St Georges Hospital, London
  - University College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - South Warwickshire Foundation Trust, Warwick

IPD SHARING:
Plan to Share IPD: No